CLINICAL TRIAL: NCT00436865
Title: Insulin and the Polycystic Ovary Syndrome
Brief Title: Insulin and the Polycystic Ovary Syndrome--Weight Reduction Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HM10313; K23HD049454-01A2 (NIH)
Record Dates: First submitted 2007-02-15; First posted 2007-02-19 (Estimated); Last update posted 2018-03-30 (Actual); Status verified 2018-03

CONDITIONS: Polycystic Ovary Syndrome; Obesity
MeSH Terms: conditions — Polycystic Ovary Syndrome; Obesity

ARMS (2):
- PCOS (Other): PCOS women receiving weight loss intervention
  Interventions: Behavioral: Weight loss
- Control (Other): Non-PCOS women receiving weight loss intervention
  Interventions: Behavioral: Weight loss

INTERVENTIONS:
Behavioral: Weight loss

SUMMARY:
The polycystic ovary syndrome is the leading cause of female infertility in the United States. The disorder affects approximately 6-10% of women of reproductive age. It is widely accepted that "insulin resistance" may be responsible for the infertility of this syndrome. Women are insulin resistant when their bodies do not respond to insulin's action to handle sugar as they normally should. Because of this insulin resistance, women with the polycystic ovary syndrome are also at high risk for developing type 2 diabetes. We have previously shown that D-chiro-inositol (DCI), a substance naturally found in our body that helps insulin's action, is lacking in women with the polycystic ovary syndrome. Not having enough DCI may lead to insulin resistance. The purpose of this study is to determine if weight loss helps to replenish the body with DCI and help to promote insulin's action.

DETAILED DESCRIPTION:
Insulin resistance is present in women with PCOS. Women with PCOS are at high risk for developing type 2 diabetes, presumably due to the insulin resistance that accompanies the syndrome. Some actions of insulin may be effected by putative inositolphosphoglycan (IPG) mediators of insulin action, and evidence suggests that a deficiency in a specific D-chiro-inositol (DCI)-containing IPG may contribute to insulin resistance in individuals with impaired glucose tolerance or type 2 diabetes mellitus. A deficiency in DCI may also contribute to the insulin resistance in women with PCOS. In PCOS, three separate studies have shown that administration of DCI, the precursor to DCI-IPG, to women with PCOS improved glucose intolerance while reducing circulating insulin, improved ovulatory function, and decreased serum androgens. Serum triglycerides, HDL cholesterol and blood pressure improved in some of the studies as well. Collectively, these findings strongly suggest that administration of DCI improved insulin sensitivity in women with PCOS, and that a deficiency in DCI may contribute to the insulin resistance of this disorder.

Previous studies of our group demonstrated that women with PCOS, when compared to normal women, had a (i) greater than 5-fold increase in the renal clearance of DCI, (ii) 50% reduction in the circulating concentration of DCI, and (iii) decreased insulin-stimulated release of DCI-IPG during an oral glucose tolerance test (OGTT). Moreover, insulin sensitivity (as determined by frequently sampled intravenous glucose tolerance test [FSIVGTT]) correlated inversely with renal clearance of DCI. In addition, it appears that obesity needs to be present for the abnormality in renal clearance of DCI to be present in PCOS, and obesity does not seem to have an effect in DCI renal clearance in normal women.

Our hypothesis is that obesity modulates the renal clearance of DCI in women with PCOS, but not in normal women. A corollary of this hypothesis is that an increased urinary DCI clearance leads to a reduction in circulating DCI and insulin-stimulated DCI-IPG release, and aggravates insulin resistance in women with PCOS. To test our hypothesis, we propose to study the following specific aims:

Specific Aims:

Specific Aim 1: Determine if DCI renal clearance in obese women with PCOS is increased compared to age- and weight-matched, obese normal women.

In this aim, we will determine if obese women with PCOS have (i) increased renal clearance of DCI, (ii) decreased circulating levels of DCI, and (iii) decreased DCI-IPG release in blood during an OGTT, as compared to age- and BMI-matched, obese normal women.

Specific Aim 2: Determine if weight loss reduces DCI renal clearance in obese women with PCOS, but not in age- and weight-matched obese normal women.

This aim determines if weight loss reverses the abnormalities in DCI handling in PCOS. The effects of weight loss on (i) renal clearance of DCI, (ii) circulating levels of DCI, and (iii) DCI-IPG release in blood during an OGTT, will be compared between obese women with PCOS and age- and BMI-matched obese normal women.

Specific Aim 3: Determine if a change (reduction) in DCI renal clearance as a result of weight loss is correlated with a change (improvement) in insulin sensitivity in obese women with PCOS that is independent of weight loss itself.

In our Preliminary Studies, we have determined that insulin sensitivity has a significant inverse relationship with urinary DCI clearance. In this aim, we will determine if decreasing DCI renal clearance by weight loss in obese women with PCOS will improve insulin sensitivity independent of the degree of weight loss (via statistical adjustment with the degree of weight loss as a covariate).

Specific Aim 4: Determine if an equivalent degree of weight loss in obese women with and without PCOS is associated with (i) a greater reduction in DCI renal clearance, and (ii) a greater improvement in insulin sensitivity in the PCOS women compared to the normal women.

To further demonstrate whether improvement in insulin sensitivity as a result of an improvement in DCI handling is independent of weight loss itself, women will be stratified by the degree of weight loss. For each degree of weight loss, we will determine if obese women with PCOS have (i) a greater reduction of renal clearance of DCI and (ii) a greater improvement in insulin sensitivity as a result of weight reduction, as compared to weight-matched obese normal women.

If our proposed studies confirm a role for obesity in modulating DCI handling in PCOS, they will substantially enhance our understanding of the pathogenesis of PCOS and are likely to provide insights into novel treatment strategies directed specifically at the IPG system and normalization of its function.

ELIGIBILITY:
Inclusion Criteria:

* Obese (≥ 30 kg/m2) premenopausal women with PCOS and normal women between 18-40 years of age.
* PCOS women only:

  * oligomenorrhea (<= 8 menstrual periods annually),
  * biochemical hyperandrogenemia (elevated total or free testosterone),
  * normal thyroid function tests and serum prolactin, and
  * exclusion of 21alpha-hydroxylase deficiency by a fasting 17alpha-hydroxyprogesterone <200 ng/dl.
* Normal women only:

  * regular monthly menses, and
  * normal serum total and free testosterone.
* All women:

  * acceptable health on the basis of interview, medical history, physical examination, and laboratory tests (CBC, SMA20, urinalysis),
  * have not been dieting in the 3 months prior to study enrollment,
  * signed, witnessed informed consent,
  * ability to comply with study requirements.

Exclusion Criteria:

* Diabetes mellitus by fasting glucose or OGTT, or clinically significant pulmonary, cardiac, renal, hepatic, neurologic, psychiatric, infectious, neoplastic and malignant disease (other than non-melanoma skin cancer).
* Documented or suspected recent (within one year) history of drug abuse or alcoholism.
* Ingestion of any investigational drug within 3 months prior to study onset.
* Pregnancy as documented by urine hCG.
* PCOS women only: Change in PCOS medication regimen (oral contraceptives, spironolactone, insulin sensitizers) within 3 months prior to the start of the study.
* Normal women only:

  * history of gestational diabetes,
  * positive family history for first-degree relative with diabetes,
  * disorders linked to insulin resistance (hypertension or dyslipidemia),
  * Use of oral or other systemic contraceptives, or spironolactone within 3 months prior to the start of the study,
  * Use of medications (including OTC drugs) known to affect insulin sensitivity such as metformin, rosiglitazone, pioglitazone, niacin, corticosteroids, beta blockers, calcium channel blockers and thiazide diuretics within 3 months prior to the start of the study.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 79 (Actual)
Dates: Start 2007-02; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Insulin sensitivity (Change from baseline to 8 weeks) | Baseline to 8 weeks
Changes of Serum D-Chiro-Inositol (DCI) concentrations (Change from baseline to 8 weeks) | Baseline to 8 weeks
Changes of DCI renal clearance (Change from baseline to 8 weeks) | Baseline to 8 weeks
Changes of AUC insulin during OGTT (Change from baseline to 8 weeks) | Baseline to 8 weeks
AUC of bioactive DCI-IPG during OGTT (Change from baseline to 8 weeks) | Baseline to 8 weeks
Ratio of AUC DCI-IPG to AUC insulin during OGTT (Change from baseline to 8 weeks) | Baseline to 8 weeks

SECONDARY OUTCOMES:
Weight loss (Change from baseline to 8 weeks) | Baseline to 8 weeks
Serum Myo-Inositol (Myo) concentrations (Change from baseline to 8 weeks) | Baseline to 8 weeks
MYO bioactivity (Change from baseline to 8 weeks) | Baseline to 8 weeks
Serum inflammatory and cardiovascular markers (Change from baseline to 8 weeks) | Baseline to 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Kai I. Cheang, Pharm.D., Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University General Clinical Research Center, Richmond, Virginia, United States